CLINICAL TRIAL: NCT00290901
Title: A Six Week Double-Blind, Randomized, Multicenter Comparison Study of the Analgesic Effectiveness of Celecoxib 200 mg BID Compared to Tramadol Hydrochloride 50 mg QID in Subjects With Chronic Low Back Pain
Brief Title: Celebrex vs Tramadol in the Treatment of Chronic Lower Back Pain.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191165
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Tramadol; Celecoxib

INTERVENTIONS:
Drug: Tramadol Hydrochloride 50mg
Drug: Celebrex 200mg

SUMMARY:
This study investigates if Celebrex is as effective as tramadol hydrochloride (Ultram) for patients with chronic low back pain, when administered over a 6-week period.

ELIGIBILITY:
Inclusion Criteria:

* The subject presents with duration of chronic low back pain of > 3 months requiring regular use of analgesics (> 4 days/week), except for acetaminophen which cannot have been the sole analgesic used.

Exclusion Criteria:

* The subject has chronic low back pain, which is neurologic in etiology (i.e., radiculopathy, neuropathy, myelopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 754
Dates: Start 2006-03; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To compare the analgesic effectiveness of celecoxib and tramadol in subjects with Chronic Low Back Pain measured by the Numerical Rating Scale (NRS-Pain) at Week 6.

SECONDARY OUTCOMES:
To compare the effects of treatment with celecoxib 200 mg BID and tramadol hydrochloride 50 mg QID on improvement in functionality and quality of life in subjects with chronic low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- United States (53):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, San Luis Obispo, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Vista, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Cos Cob, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Woodstock, Georgia
  - Pfizer Investigational Site, Libertyville, Illinois
  - Pfizer Investigational Site, Morton Grove, Illinois
  - Pfizer Investigational Site, Arkansas City, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Camp Hill, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, San Angelo, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Danville, Virginia
- Pfizer Investigational Site, Rio Piedras, Puerto Rico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191165&StudyName=Celebrex+vs+Tramadol+in+the+treatment+of+chronic+lower+back+pain%2E+